CLINICAL TRIAL: NCT04026464
Title: Monotherapy (Ibuprofen) vs. Combination Therapy (Ibuprofen and Acetaminophen) in the Management of Patent Ductus Arteriosus in Premature Infants: A Randomized Controlled Trial
Brief Title: Addition of Acetaminophen in Standard PDA Management
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain funding to support this project
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201901829 -A
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen+Acetaminophen Group (Active Comparator): Infants with PDA randomized to the combined treatment group receiving intravenous ibuprofen (10 mg/kg intravenous ibuprofen followed by 5 mg/kg 24 and 48 hours subsequently) and oral acetaminophen (15 mg/kg oral acetaminophen [160 mg/5ml concentration] every 6 hours for a total of 12 doses).
  Interventions: Drug: Intravenous Ibuprofen + Oral Acetaminophen
- Ibuprofen Group (Placebo Comparator): Infants with PDA randomized to the control mono therapy group receiving intravenous ibuprofen (10 mg/kg intravenous ibuprofen followed by 5 mg/kg 24 and 48 hours subsequently) alone.
  Interventions: Drug: Intravenous Ibuprofen

INTERVENTIONS:
Drug: Intravenous Ibuprofen — The control monotherapy group will receive 10 mg/kg intravenous ibuprofen followed by 5 mg/kg 24 and 48 hours subsequently.
  Arms: Ibuprofen Group
Drug: Intravenous Ibuprofen + Oral Acetaminophen — The combined treatment group will receive 10 mg/kg intravenous ibuprofen followed by 5 mg/kg 24 and 48 hours subsequently and will in addition receive 15 mg/kg oral acetaminophen [160 mg/5ml concentration] every 6 hours for a total of 12 doses.
  Arms: Ibuprofen+Acetaminophen Group

SUMMARY:
Patent ductus arteriosus is a common morbidity in preterm infants and management of PDA varies among neonatologist. The investigators are conducting a randomized controlled trial to determine the rates of initial patent ductus arteriosus (PDA) closure after completion of a first treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Infants 23 0/7 to 27 6/7 weeks' gestational age and birth weight < 1000 grams
* Hemodynamically significant PDA as defined by any of the following:

  1. Increased ventilator or oxygen support attributed by the clinician to be due to increased left-right shunting through the PDA
  2. Hypotension and/or widening pulse pressure requiring continuous dopamine infusion (hypotension is defined as mean arterial pressure (MAP) at least 2-3 mmHg below the infants' post menstrual age)
  3. Signs of congestive heart failure (e.g increased pulmonary congestion on chest radiograph or hepatomegaly on physical examination)
* Echocardiographic criteria:

  1. Ratio of the smallest ductal diameter to the ostium of the left pulmonary artery > 0.5

Exclusion Criteria:

* No enteral feedings
* PDA-dependent congenital heart disease
* Prior treatment with prophylactic indomethacin
* Prior PDA treatment with any medications
* Suspected or diagnosed acute necrotizing enterocolitis (NEC) or spontaneous intestinal perforation
* Abnormal liver enzymes (ALT > 60 IU/L and AST > 60 IU/L)
* Platelets count < 50,000 /μl; and / or active intracranial, gastrointestinal, or other bleeding
* Major congenital anomalies such as neural tube defect, known or suspected chromosomal abnormality, and gastrointestinal defect
* Prior enrollment to other interventional clinical study where PDA is an outcome variable

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Percentage of infants with PDA closure. | During hospitalization, up to 10 days
  Percentage of patients who demonstrated PDA closure.

CONTACTS AND LOCATIONS:
Overall Officials: Sanket D Shah, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No